CLINICAL TRIAL: NCT07120646
Title: The Co-Morbidity of Pain and Sleep Disturbances in Children Living Beyond Cancer: A Case-Control Study
Brief Title: Pain and Sleep Disturbances in Children Living Beyond Cancer: A Case-Control Study
Status: Not yet recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Emma Rheel, Dr., Vrije Universiteit Brussel
Other Study IDs: PEEPTrial_CaseControl
Record Dates: First submitted 2025-06-26; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Childhood Cancer Survivors
Keywords: children living beyond cancer; pain; sleep disturbances; case-control
MeSH Terms: conditions — Pain; Parasomnias | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children living beyond cancer (CBC)
  Interventions: Other: Questionnaire, actigraphy measurement and sleep diary
- healthy controls: age- and sex-matched healthy controls
  Interventions: Other: Questionnaire, actigraphy measurement and sleep diary

INTERVENTIONS:
Other: Questionnaire, actigraphy measurement and sleep diary — Baseline questionnaires (measuring socio-demographic and health-related information, as well as most outcome measures), followed by 2 weeks of actigraphy measurement and daily sleep diary.

SUMMARY:
Children living beyond cancer (CBC) represent a unique and growing population of young people in need of long-term clinical support. Studies suggest that 11-44% of CBC experience chronic pain, negatively impacting a wide range of child biopsychosocial outcomes and creating high financial burden for their families and society. Often comorbid with pain, one of the most chronic and disturbing side effects reported by CBC are sleep disturbances, and in particular, difficulties initiating and maintaining sleep. Indeed, >50% of CBC report some form of sleep disturbance even 9 to 15 years after the cancer diagnosis. Much attention has been paid to sleep and pain as independent constructs within pediatric oncology, yet Belgian data is lacking. Additionally, little is known about how these domains interact with one another and subsequent indications for prevention and intervention. Although evidence shows an interrelationship between pain and sleep in adult and pediatric populations, this interrelationship is understudied in childhood cancer patients and CBC. (Chronic) pain may serve as a modifiable target for interventions to improve sleep quality and vice versa, and understanding this relationship is crucial for providing comprehensive care to CBC. Therefore, this cross-sectional case-control study aims to explore the differences in pain and sleep disturbances in CBC compared to healthy age- and sex-matched healthy controls, as well as the interrelationship between both outcomes.

DETAILED DESCRIPTION:
Pain and sleep disturbances are common and impactful following childhood cancer treatment

Worldwide, about 400 000 children aged 0-19 years are diagnosed with cancer each year. Largely due to more intensive treatment regimens and the implementation of immunotherapy for high-risk patients, 5-year survival rates for children with cancer in high income countries have increased to >80%. This is great news, however as a result, children living beyond cancer (CBC) represent a unique and growing population of young people in need of long-term clinical support.

Across the cancer continuum, pain is a prevalent, recurrent, and impactful symptom. Although we know that pain in childhood cancer is underreported and undertreated, the prevalence of pain in children during active cancer treatment varies from 28-62% across studies, with >50% of children reporting moderate to severe pain intensity. For many children, pain resolves following completion of the cancer treatment, yet for some, pain persists well beyond treatment7 and into adulthood. Indeed, studies suggest that 11-44% of CBC experience chronic pain (i.e., pain in ≥ 1 anatomic region persisting or recurring for >3 months), with 20% reporting moderate to extreme pain interference. Chronic pain can deleteriously impact the lives of CBC and their family. Specifically, if not addressed early on, chronic pain can negatively impact children's school functioning, sleep quality, social and family functioning, mental health, physical activity, and overall health-related quality of life. Moreover, it increases the risk of chronic pain across the lifespan. Further, also the families of children with chronic pain can experience significant physical and psychosocial sequelae due to the child's pain, e.g., high levels of anxiety and depressive symptoms, and a high financial burden due to direct and indirect medical costs.

Often comorbid with pain, one of the most chronic and disturbing side effects reported by childhood cancer patients and CBC are sleep disturbances, and in particular, difficulties initiating and maintaining sleep, suggesting that this is a major quality of life concern. Indeed, >50% of CBC report some form of sleep disturbance even 9 to 15 years after the cancer diagnosis. Good-quality sleep in childhood is crucial for a healthy emotional, cognitive, physical, and behavioral development. Healthy sleep involves receiving a developmentally appropriate number of hours of sleep (declining from infancy to adolescence), few or preferably no wakings during the night, and a subjective perception of feeling rested. CBC may be at increased risk for sleep disturbances, being critically ill during a life phase that is important in the development of good sleep habits. Disrupted sleep can also affect inflammatory pathways and immune functioning, incl. natural killer cell activity, and can contribute to or exacerbate other morbidities common to survivorship (e.g., anxiety, depression). Sleep disruption is unlikely to remit without intervention and longitudinal research shows that sleep disruption often persists from childhood into adolescence.

Study Rationale and Purpose

Some attention has been paid to sleep and pain as independent constructs within pediatric oncology, although Belgian data is lacking and little is known about how these domains interact with one another and subsequent indications for prevention and intervention. Early studies propose a bi-directional relationship between pain and sleep, such that sleep deficiency and pain reciprocally maintain symptoms over time. Yet, the interrelationship between pain and sleep is understudied in childhood cancer patients and CBC. (Chronic) pain may serve as a modifiable target for interventions to improve sleep quality and vice versa, and understanding this relationship is crucial for providing comprehensive care to CBC.

This cross-sectional case-control study aims to explore the differences in pain and sleep disturbances in CBC (6-12 years old) compared to healthy age- and sex-matched healthy controls, as well as the interrelationship between both outcomes.

ELIGIBILITY:
Inclusion Criteria:

* CBC: 1) current age 6-12yo; 2) history of any cancer diagnosis; 3) ≤ 5y post- treatment completion; 4) ≥ 3 months since last cancer treatment (since pain and insomnia during treatment can be directly related to therapy and recover spontaneously); 5) fluent Dutch speaker and reader (age-dependent)
* Healthy controls (age- and sex-matched): 1) current age 6-12yo; 2) no history of cancer ; 3) fluent Dutch speaker and reader (age-dependent)
* Parents: 1) fluent Dutch speaker and reader

Exclusion Criteria:

* CBC: 1) receiving palliative therapy; 2) psychiatric disorder; 3) severe intellectual disability
* Healthy controls: 1) history of cancer; 2) psychiatric disorder; 3) severe intellectual disability

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children living beyond cancer (6-12 years old) and age- and sex-matched healthy controls, together with one of their parents.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Activity limitations due to pain | Baseline about the past 14 days + 14 days following baseline in daily sleep diary
  Measured with the Child Activity Limitations Interview (CALI) - 9 (parent-report version for the 6-7 year-olds; self-report version for the 8-12 year-olds)
Sleep disturbances | Baseline
  Assessed with the PROMIS Parent Proxy Item Bank v1.0 - Sleep Disturbance - Short Form 8a parent-report for the 6-7 year olds and PROMIS Pediatric Item Bank v1.0 - Sleep Disturbance - Short Form 8a for the 8-12 year-olds. Additionally, this outcome measure is assessed with the Children's Sleep Habits Questionnaire (CSHQ) (parent-report for all ages).

SECONDARY OUTCOMES:
Pain severity | Baseline
  Assessed with the Pain Frequency Severity Duration scale (PFSD) (parent-report for the 6-7 year-olds; self-report for the 8-12 year-olds)
Pain coping | Baseline
  Assessed with the Pain Coping Questionnaire short form (parent-report for the 6-7 year-olds; self-report for the 8-12 year-olds)
Pain reporting and assessment during follow-up care | Baseline
  Assessed using a selfmade set of items about pain reporting and assessment during medical follow-up consultations
Health-related quality of life | Baseline
  Assessed with the PedsQL Generic Score Scales 4.0 (5-7yo parent-report) for the 6-7 year-olds and the PedsQL Generic Score Scales 4.0 (8-12yo self-report) for the 8-12 year-olds.
Fatigue | Baseline
  Assessed with the PedsQL Multidimensional Fatigue Scale 3.0 (5-7yo parent-report) for the 6-7 year-olds and the PedsQL Multidimensional Fatigue Scale 3.0 (8-12yo self-report) for the 8-12 year-olds.
Anxiety | Baseline
  Assessed with the PROMIS Parent Proxy 3.0 - Anxiety - Short Form 8a for 6-7 year-olds and the PROMIS Pediatric 3.0 - Anxiety - Short Form 8a for the 8-12 year-olds.
Depressive symptoms | Baseline
  Assessed with the PROMIS Parent Proxy 3.0 - Depressive Symptoms - Short Form 6a for the 6-7 year-olds and the PROMIS Pediatric 3.0 - Depressive Symptoms - Short Form 6a for the 8-12 year-olds.
Total sleep time | 14 days following baseline
  The total amount of time scored as sleep in minutes from sleep onset to sleep offset. Assessed with Actigraphy (Fitbit Sense 2)
Wake minutes after sleep onset | 14 days following baseline
  The number of minutes scored as wake after nighttime sleep onset. Assessed with Actigraphy (Fitbit Sense 2)
Sleep efficiency | 14 days following baseline
  The ratio of total sleep time and total time spent in bed at night as a percentage, with values closer to 100 indicating more efficient sleep. Assessed with Actigraphy (Fitbit Sense 2)
Sleep regularity index | 14 days following baseline
  Similarity of the child's sleep-wake pattern from one day to the next based on binary sleep-wake time series. Assessed with Actigraphy (Fitbit Sense 2)
Pain symptoms during the day | 14 days following baseline
  This data is collected via a daily sleep diary and includes: presence of pain (yes/no), and if yes; mean and worst pain during the day (0 = no pain; 10 = worst pain possible)
Medication intake during the day | 14 days following baseline
  This data is collected via a daily sleep diary and includes whether the child took medication during the day (yes/no), and if yes; which medication.

OTHER OUTCOMES:
Information about prior night's sleep pattern and day | From baseline to 14 days later
  This data is collected via a daily sleep diary to interpret the Actigraphy data (bedtime, time of falling a sleep, number of wakings during the night, time of waking up in the morning, time of getting up in the morning, time and reasons for taking of the Fitbit, time of naps)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Rheel, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be documented both at the project level and at the data level:
  Data level:
  * In research papers;
  * Information about variables using labels and variables derivations
  Project level
  * Documentation about the authors, background, aims, objectives, and the hypotheses that shape the research
  * Data collection protocol & procedures
  * Project meeting reports
  Descriptive metadata of data items will be registered in Pure Database with restricted acces (closed access, only on reasonable request). In addition, the raw dataset will include labels in the .xlsx file including variable information providing documentation at the data level. Datasets will be accompanied by a separate word.doc file providing study-level documentation including the field methods used for data collection.
Time Frame: Within one year following the end of the study, for 10 years.
Access Criteria: Closed access (only on reasonable request)
URL: https://dmponline.be/